CLINICAL TRIAL: NCT07246174
Title: Comparison of AH Plus and WellRootST Root Canal Sealers in Terms of Postoperative Pain: One-Month Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Furkan Salih Bilgi, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-243
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Root Canal Treatment
Keywords: epoxy-resin-based root canal sealers; Calcium silicate-based root canal sealer; postoperative pain; Visual Analog Scale
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AhPlus sealer (Experimental): AH Plus sealer used
  Interventions: Procedure: AH-Plus Epoxy Resin Sealer
- WellRootST sealer (Experimental): WellRootST sealer used
  Interventions: Procedure: bioceramic sealer

INTERVENTIONS:
Procedure: AH-Plus Epoxy Resin Sealer — AhPlus sealer was used for group 1
  Arms: AhPlus sealer
Procedure: bioceramic sealer — WellRootSt wa used for group 2
  Arms: WellRootST sealer

SUMMARY:
The objective of this research was to identify which of the root canal sealers, AH Plus or WellRootST, yielded more effective outcomes regarding postoperative pain when applied to teeth diagnosed with apical periodontitis.

DETAILED DESCRIPTION:
A prospective cohort study was conducted at a single center, involving 120 patients diagnosed with chronic apical periodontitis (AP) admitted for endodontic treatment. Patients were categorized into two groups based on the type of root canal sealer used. Sixty patients treated with AH Plus sealer constituted Group 1, while sixty patients treated with WellRootST sealer comprised Group 2. Data collected for all participants included age, gender, findings from oral and dental examinations, tooth type, tooth number, duration of root canal treatment, and Visual Analog Scale (VAS) results recorded preoperatively, as well as at 24 hours, 48 hours, 72 hours, 1 week, and 1 month postoperatively.

ELIGIBILITY:
The inclusion criteria for this study were as follows:

1. Participants had to be at least 18 years old
2. One mature tooth showing signs or symptoms that required primary root canal treatment.
3. Participants needed to be in good general health
4. classified as ASA I or II, and able to follow the follow-up schedule.

Exclusion criteria criteria for this study were as follows:

1. Included teeth with internal or external root resorption,
2. Signs of perforation
3. The need for post-core application, or previous restoration with fixed prosthetic appliances, such as crowns or bridges

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative pain evaluation by VAS scale | Baseline, 24 hour postoperatively, 48hour postoperatively, 72 hour postoperatively, Day 3 and Day 7
  Study groups were compared in terms of VAS scores at the preoperative period and postoperative 24 hours, 48 hours, 72 hours, 1 week, and 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Furkan S Bilgi, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Upon request from the authors with a reasonable request, our data will be made open
Supporting Information: Study Protocol, SAP
Time Frame: After the acceptance of our study
Access Criteria: Our data will be shared via email